CLINICAL TRIAL: NCT03253328
Title: N-Acetyl-Cysteine for Healing of Amputation Stumps in the Setting of Diabetes
Brief Title: N-Acetyl-Cysteine (NAC) for Healing of Amputation Stumps in the Setting of Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201611065
Record Dates: First submitted 2017-03-17; First posted 2017-08-17 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus; Critical Limb Ischemia; Lower Limb Amputation Knee; Peripheral Arterial Disease
MeSH Terms: conditions — Diabetes Mellitus; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Arm N-acetyl cysteine (NAC) (Active Comparator): Upon study enrollment, patients will be randomized 1:1 by Investigational Pharmacy to a standard adult intravenous dose of NAC (1200mg twice a day) for 6 days post-amputation.
  Interventions: Drug: Active Arm N-acetyl cysteine (NAC)
- Placebo Arm (Placebo Comparator): Upon study enrollment, patients will be randomized 1:1 by Investigational Pharmacy to placebo ½ normal saline infusion (twice a day) for 6 days post-amputation.
  Interventions: Drug: Placebo Arm

INTERVENTIONS:
Drug: Active Arm N-acetyl cysteine (NAC) — N-acetyl cysteine (NAC) 1200mg twice a day for 6 days post-amputation
  Other Names: N-acetyl cysteine (NAC)
  Arms: Active Arm N-acetyl cysteine (NAC)
Drug: Placebo Arm — Placebo 1/2 normal saline infusion twice a day for 6 days post-amputation
  Other Names: Placebo 1/2 normal saline infusion
  Arms: Placebo Arm

SUMMARY:
In this pilot clinical study the investigators propose to conduct a prospective, randomized, double-blinded, placebo-controlled clinical trial for 30 days for participants with critical limb ischemia (CLI) who undergo a major (above-knee or below-knee) lower extremity amputation. By exploring the primary endpoints we aim to determine whether NAC can affect amputation stump perfusion and healing. Based on preclinical data, the investigators hypothesize that NAC will augment both amputation stump perfusion as well as healing. The investigators will utilize the data from this trial to determine the true effect size that is necessary for a larger clinical trial to determine the clinical efficacy of NAC is healing surgical sites such as major lower extremity amputation stumps.

DETAILED DESCRIPTION:
In this pilot clinical study the investigators propose to conduct a prospective, randomized, double-blinded, placebo-controlled clinical trial, in 50 participants with CLI who have undergone a major (above-knee or below-knee) lower extremity amputation. 25 participants will receive NAC 1200mg intravenously twice a day for 6 consecutive days following amputation. 25 participants will receive placebo saline intravenous infusion twice a day for 6 days following amputation. Post-amputation participants will be monitored for specific anthropometric parameters and stump perfusion assessments (using laser-assisted fluorescent angiography and transcutaneous oxygen pressure measurement). The primary study endpoints are to determine if lower extremity stump healing and perfusion are affected by perioperative NAC administration. A secondary endpoint will be to determine the effect size that would be necessary to power a larger clinical trial to determine whether NAC treatment can affect tissue perfusion and healing at major lower extremity amputation stumps in participants with CLI.

ELIGIBILITY:
Inclusion Criteria:

* Subject undergoing elective major (above-knee or below-knee) lower extremity amputation for CLI
* Both male and female patients
* All ethnic groups
* Between of the ages of 30-90 years old
* Adequate nutritional status - defined as BMI > 19

Exclusion Criteria:

* Pregnant women, and women who are breastfeeding
* Known history of end-stage liver disease
* Severe asthma
* Heavy alcohol consumption (male > 2 drinks per day and women > 1 drink per day)
* Individuals actively receiving chemotherapy.
* Anticipated enrollment in another study that investigates another drug agent within 30 days from enrollment in this study.
* Patients receiving carbamazepine.
* Severe anemia (HCT < 22).
* Allergy to either NAC or Indocyanine Green (ICG).
* Patients with open wound(s) from a prior amputation on the ipsilateral limb (excluding patients who had prior partial foot amputation, who are now requiring a below-knee or above-knee amputation).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zayed, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JV, Engel C, Tay S, DeSilva G, Desai K, Cashin J, Semenkovich CF, Zayed MA. Impact of N-Acetyl-Cysteine on Ischemic Stumps Following Major Lower Extremity Amputation: A Pilot Randomized Clinical Trial. Ann Surg. 2022 Nov 1;276(5):e302-e310. doi: 10.1097/SLA.0000000000005389. Epub 2022 Jan 24. PMID 35129469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from March 2017 to April 2020. We initially planned to enroll 15 subjects in each group but recruitment was suspended in May 2020 due to COVID-19. Study team leadership determined that unmasking of study randomization would facilitate analysis of primary/secondary endpoints and determine whether data supported overall study hypothesis. After pandemic disruptions were eased interim study analysis was completed and the study closed. No safety concerns led to early termination.
Period: Overall Study
Arm/Group | Active Arm N-acetyl Cysteine (NAC) | Placebo Arm
Started | 16 | 17
Completed | 10 | 16
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm N-acetyl Cysteine (NAC) | Placebo Arm | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Median (Standard Deviation); unit: years] | 69 (12) | 62 (11) | 65.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Postoperative Laser-Assisted Fluorescent Angiography (LAFA) Perfusion.
Description: Images were collected from the SPY Elite LAFA apparatus. Regions of interest were drawn in a standardized fashion around either the incision or the whole amputation stump. NIH image J software was used to evaluate peak perfusion signal intensity in all regions of interest. Change in LAFA was assessed at postoperative day (POD) 0, 3, and 5. Fold change in % perfusion in the ROI's between POD 0/3/5 was determined and compared between study groups. The primary outcomes were change in postoperative Laser-Assisted Fluorescent Angiography (LAFA) perfusion at POD3 and POD5 and stump healing at postoperative day 30 (POD30).
Time Frame: Day 0, Day 3, Day 5
Population: Table represents fold change in amputation stump % perfusion defect between POD 0, 3, 5.
Measure: Mean (Standard Deviation); unit: percentage of defect
Arm/Group | Active Arm N-acetyl Cysteine (NAC) | Placebo Arm
Number analyzed (Participants) | 10 | 16
percentage of defect
  POD 0: number analyzed (Participants) | 7 | 13
  POD 0 | 0.060 (0.056) | 0.096 (0.117)
  POD 3: number analyzed (Participants) | 7 | 13
  POD 3 | 0.045 (0.047) | 0.031 (0.055)
  POD 5: number analyzed (Participants) | 7 | 13
  POD 5 | 0.015 (0.026) | 0.050 (0.058)

2. Primary Outcome: Stump Healing Assessment at Postoperative Day (POD) 30.
Description: Amputation stump photographs were serially obtained for all study patients immediately before LAFA assessments on POD 0, 3, and 5. A blinded observer evaluated amputation stump incision healing using a modified Bates-Jensen Score (mBJS) wound assessment tool. As previously described, the amputation stumps were evaluated on the following criteria: amputation stump skin color, epithelialization, amount of exudate, and the presence and volume of eschar. Each wound healing characteristic was given a score of 1 to 5, with higher scores indicating worse healing. Eschar volume was determined using ImageJ software. Aggregate mBJS scores were derived for both the whole stump and along the suture line. Clinical amputation stump healing was determined by the surgeon at follow-up clinical evaluations up until POD30.
  De Silva GS, Saffaf K, Sanchez LA, et al. Amputation stump perfusion is predictive of post-operative necrotic eschar formation. Am J Surg. 2018;216:540-546.
Time Frame: 30 days
Population: Amputation Stump Incision Healing
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm N-acetyl Cysteine (NAC) | Placebo Arm
Number analyzed (Participants) | 10 | 16
Participants
  Overall Number of Participants Analyzed | 10 | 16
  Perfusion Defects | 7 | 13
  Adequate Perfusion | 3 | 3

3. Secondary Outcome: Amputation Stump Perfusion in High Risk Patients
Description: POD0 LAFA was evaluated for all patients and patients that demonstrated amputation stump peak perfusion defects were considered high risk. Within these patients we then evaluated amputation stump perfusion at POD5.
  Change in perfusion over this time was compared between the study groups.
Time Frame: POD5
Population: Amputation stump perfusion at POD5.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm N-acetyl Cysteine (NAC) | Placebo Arm
Number analyzed (Participants) | 10 | 16
Participants
  Perfusion Defects | 7 | 13
  Adequate Perfusion | 3 | 3

ADVERSE EVENTS:
Time Frame: Postoperative Day 30 (POD30)
Description: There were no study-related adverse events observed throughout the duration of this clinical trial.
Groups:
- PLACEBO: Upon study enrollment, patients will be randomized 1:1 by Investigational Pharmacy to placebo ½ normal saline infusion (twice a day) for 6 days post-amputation.
  Placebo Arm: Placebo 1/2 normal saline infusion twice a day for 6 days post-amputation
Arm/Group | Active Arm N-acetyl Cysteine (NAC) | PLACEBO
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 6/16 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm N-acetyl Cysteine (NAC) (N=16) | PLACEBO (N=17)
Non-healing amputation site (Vascular disorders) | 1 (1) | 0 (0) — Non-healing amputation site
Conversion from BKA to AKA (Surgical and medical procedures) | 0 (0) | 1 (1) — Conversion from below knee amputation (BKA) to above knee amputation (AKA)
Erosive esophagitis (General disorders) | 1 (1) | 0 (0) — Erosive esophagitis
Stump pain (Vascular disorders) | 0 (0) | 1 (1) — Stump pain
Constipation resulting in hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Constipation resulting in hospitalization
Fecal impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Fecal impaction
Wound necrosis (Infections and infestations) | 0 (0) | 1 (1) — Wound necrosis
Hypovolemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Hypovolemia
Diabetic ketoacidosis (DKA) (Endocrine disorders) | 1 (1) | 0 (0) — Diabetic ketoacidosis (DKA)
Amputation stump revision due to a fall (General disorders) | 1 (1) | 0 (0) — Amputation stump revision due to a fall
Death (Infections and infestations) | 1 (1) | 0 (0) — Complications associated with diabetic ketoacidosis (DKA)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03253328/Prot_SAP_ICF_000.pdf